CLINICAL TRIAL: NCT00584402
Title: Contrast Sonography for Evaluation of Liver Tumors Prior to Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200715241
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Liver Neoplasms
Keywords: liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast sonography (Experimental): Contrast-enhanced sonography perflutren lipid microspheres
  Interventions: Drug: perflutren lipid microspheres

INTERVENTIONS:
Drug: perflutren lipid microspheres — perflutren lipid microspheres IV in 0.1 cc doses, as needed, to enhance lesion conspicuity
  Other Names: Definity

SUMMARY:
The purpose of this study is to determine the efficacy of the Definity (perflutren lipid microsphere Injectable Suspension) ultrasound contrast agent in identifying small tumors (hepatomas & metastases) within the liver.

Primary objective: To estimate the increase in conspicuity of small intrahepatic tumors with contrast-enhanced sonography

Secondary Objectives: To estimate the effect of tumor type, size, location and depth on the conspicuity of small tumors on contrast-enhanced sonography

DETAILED DESCRIPTION:
An estimated 75 patients (age 18 years of age or older) will be enrolled from the population of patients who present for ultrasound-guided radiofrequency ablation (RFA) of CT or MRI-confirmed multiple primary hepatocellular carcinoma (HCC) or metastatic carcinoma, with at least one of the tumors being ≤ 1.5 cm in diameter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hepatocellular carcinoma (HCC) or secondary (metastatic) carcinoma of the liver who have been referred for ultrasound-guided radiofrequency ablation (RFA) treatment
* Recent (within 90 days) CT or MRI scan with report of one or more tumors ≤ 1.5 cm in diameter
* Patient is stable and is to be managed conservatively (i.e. non-surgically)
* 18 years of age or older
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Known or suspected cardiac shunt(s)
* Known sensitivity to octafluoropropane
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. McGahan, M.D., Principal Investigator — UC Davis School of Medicine Dept. of Radiology
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Closed to enrollment
Pre-assignment Details: Closed to enrollment
Groups:
- Contrast Sonography: Contrast-enhanced sonography
  perflutren lipid microspheres : IV in 0.1 cc doses, as needed, to enhance lesion conspicuity
Period: Overall Study
Arm/Group | Contrast Sonography
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Contrast Sonography
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 5
  Female | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent of Tumors With Increased Echogenicity (Brightness) Following Contrast-enhanced Sonography
Description: After the systemic iv injection of ultrasound contrast, the real time ultrasound images are visually evaluated, and small intrahepatic tumors are detected on the images. The images pre-contrast and post contrast are compared visually. One tumor per participant was analyzed.
Time Frame: 15 min
Population: Tumors were evaluated prior and post contrast injection, 1 tumor per participant
Measure: Count of Units; unit: tumor
Units Other Than Participants: tumor
Groups:
- Contrast Sonography: Subjects undergoing contrast sonography
Arm/Group | Contrast Sonography
Number analyzed (Participants) | 8
Number analyzed (tumor) | 8
tumor | 8

2. Secondary Outcome: Number of Participants With an Increase in Echogenicity (Brightness) of Small Intrahepatic Tumors Following Contrast-enhanced Sonography Based on Tumor Type, Size, Location and Depth
Description: Visual estimation of the the effect of tumor type, size, location and depth on the conspicuity of small tumors on contrast-enhanced sonography using prior assessment or pathology for tumor type
Time Frame: 15 min
Population: Tumor types showed differences in enhancement
Measure: Number; unit: participants
Arm/Group | Contrast Sonography
Number analyzed (Participants) | 8
participants | 8

ADVERSE EVENTS:
Time Frame: 15 min post injection
Description: All-cause mortality and other (not including serious) adverse events were not collected/assessed
Arm/Group | Contrast Sonography
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less